CLINICAL TRIAL: NCT02113371
Title: Creating Health and Safety Communities of Practice for Home Care Workers
Brief Title: Evaluation of COMmunity of Practice And Safety Support (COMPASS) for Home Care Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ryan Olson, Scientist, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: e5473; U19OH010154-01 (NIH); U19OH010154-02 (NIH)
Record Dates: First submitted 2014-03-11; First posted 2014-04-14 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Wounds and Injuries; Health Promotion
Keywords: Injury Prevention; Health Promotion; Well being; Safety; Nutrition; Physical Activity; Sleep; Stress
MeSH Terms: conditions — Wounds and Injuries; Motor Activity | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention consists of monthly scripted, peer-led social support sessions covering health and safety topics.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Usual practices with regard to health and work conditions.

INTERVENTIONS:
Behavioral: Intervention
  Arms: Intervention

SUMMARY:
The current project is a safety and health intervention for home care workers conducted within the Oregon Healthy Workforce Center (OHWC), a NIOSH Center of Excellence in Total Worker Health.

The objective of this five-year project is to create sustainable health and safety "communities of practice" within a population of typically isolated home care workers. The intervention is a team-based, peer-led scripted curriculum that integrates health promotion and protection topics, as well as proven elements of social support groups for caregivers. The investigators hypothesize that this intervention will increase measures of experienced community of practice, well-being, and diet, exercise, and safety behaviors, as compared to a usual practices control condition.

DETAILED DESCRIPTION:
Home care workers have an injury rate that is nearly four times higher than the US average and are at elevated risk for mental and physical health problems. These low income workers, who are predominantly female and older than 40, assist the elderly and disabled with self-care and mobility in private homes. Although interventions developed for other caregiver populations improve well being and knowledge, they have largely failed to address illness and injury prevention behaviors. No prior study has addressed the lack of occupational social support structures for home care workers. The long term goal of this project is to create a model work structure for promoting and protecting home care worker health that can be disseminated to other states. The objective of this study is to develop and evaluate a new team-based intervention for self-employed home care workers enrolled in Oregon public programs. Workers will be organized into neighborhood based Total Worker Health teams that meet regularly for education and social support. The proposed curriculum will integrate health promotion and protection topics, and will use established team-based education methods as well as proven elements of social support groups for caregivers.

The primary hypotheses are that organizing home care workers into Total Worker Health teams will increase (1) Experienced community of practice, (2) Well-being, and (3) Prevention behaviors in the domains of diet, exercise, and safety.

The project will be conducted over five years and accomplish six specific aims. Aims 1-3 will be assessed during years 1-3, and aims 4-6 will take place during years 4 and 5.

1. Develop and Pilot Test a Total Worker Health Team Curriculum for Home Care Workers During the first year of the project the investigators will develop and pilot test a Total Worker Health team curriculum with a single group of home care workers identified as leaders by the Service Employees International Union (SEIU Local 503). Pilot test participants will later serve as team leaders in the randomized controlled trial in Aim 2. Curriculum materials will include educational workbooks, active home work assignments, and scripted meeting facilitation guides for team leaders. The curriculum will be designed to establish functioning Total Worker Health teams in 6 months using a half-day team building orientation followed by structured monthly educational and supportive team meetings. Study methods will be evaluated and revised based on pilot participants' feedback about the acceptability of the goals, procedures, and outcomes of intervention activities.
2. Determine the Effectiveness of Total Worker Health Teams with a Randomized Controlled Trial The investigators will recruit a sample home care workers from the Portland and Eugene metro areas. This sample will then be organized into neighborhood clusters and randomly assigned to intervention and control conditions. Evaluation measures will be collected from all participants at pre-intervention (month 0), post-intervention (month 6), and follow-up (month 12) time points. Intervention participants will complete the Total Worker Health curriculum while control participants receive usual treatment. Intervention effectiveness will be established at the 6-month time point through between group comparisons on changes in experienced community of practice, well-being, and prevention behaviors (diet, exercise, and safety). The investigators will also measure body composition and fitness, metabolic and heart disease biomarkers, job stress, social support, musculoskeletal symptoms, and illness/injuries.
3. Measure the Integrity of Sustained Total Worker Health Team Meetings and Maintenance at Follow-Up. After each Total Worker Health team completes the intervention curriculum, they will be provided with additional meeting topics and funding to sustain regular team meetings for an extra 6 months. The researchers will observe and monitor team meetings during this follow-up period to measure participation level and adherence to the prescribed team meeting structure. The integrity scores for team meetings and potential maintenance of between group intervention effects will be evaluated at the 12-month (follow up) time point.
4. Measure the Durability and Economic Impact of Intervention Effects and the Social Experiences of Program Participants, Within our Original Cohort. The researchers will conduct additional follow-up data collection with our original cohort at the 24-month time point to assess post-intervention maintenance. The economic impact of the intervention will be measured by computing intervention costs and contrasting them with estimated outcome-related savings for stakeholders. A qualitative study of co-worker social support within the intervention will also be implemented as part of Aim 4.
5. Adapt and Assess the Intervention for Statewide Dissemination. The intervention will be adapted for use in the existing Oregon Home Care Commission (OHCC) training system. The OHCC is the state-based employer of record for bargaining with the SEIU Local 503 and has a strong training program that reaches approximately 60% of home care workers in the state. The investigators will work with stakeholders to adapt the 12-month, 1 meeting per month Total Worker Health intervention curriculum to an accelerated 3.5-month, 2 meeting per month edition. The adapted intervention will then be assessed using a pre/post design in Oregon cities with high training attendance records using observational and selected survey outcome measures from the original randomized trial. Promotional products and resources will also be created in year 5 to support the dissemination of the adapted intervention within the OHCC and beyond.
6. Develop Relationships and Preliminary Data to Guide Translation and Dissemination With Private Agencies. The investigators will engage with private home care agencies and conduct qualitative research with agency leaders and employees to understand their organization, culture, and drivers related to the adoption of a Total Worker Health program. To do this the researchers will attend quarterly meetings of the Oregon Health Care Association, an organization which facilitates meetings with private home care agency owners from around the state. From these meetings the investigators will recruit a sample of agency and regional leaders to take part in survey completion and key informant interviews. Interviews and survey data collection with home care workers employed at several private home care agencies will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Currently employed as a home care worker with a minimum of one consumer employer

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2011-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in experienced community of practice at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Survey measures: Experienced Community of Practice Scale (Cadiz, Sawyer & Griffith, 2009).
Change from baseline in well-being at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Survey measures: SF-12 version 2 (Ware et al., 2002), Center for Epidemiologic Studies Depression Scale (CES-D) (Bohannon et al., 2003), Loneliness (Hughes et al., 2008), Positive and Negative Affect (Watson et al., 1988).
Change from baseline in dietary behaviors at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Survey measures: National Cancer Institute Fruit and Vegetable Screener (Thompson et al., 2002), High-Saturated Fat/High-Sugar Food Servings (Buxton et al., 2009).
Change from baseline in exercise behaviors at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Survey measures: Healthy physical activities scale (Elliot et al., 2007).
Change from baseline in safety behavior counts at 6 and 12 months, Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Survey measures: Reports of the frequency of safety actions (items created for the study) addressing tools/techniques for material and client moving tasks, tools/techniques for housekeeping tasks, correcting slip/trip fall hazards in homes, correcting other safety hazards, and safety communication. All items were assessed on the same frequency count scale of 0 to 5+ occurrences in the past six months.
Change from baseline safety behavior consistency at 6 and 12 months, Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Survey measures: Reports of the frequency of safety actions (items created for the study) addressing safe tools or techniques for client moving or transferring tasks, moving or lifting objects, assisting a client with walking, working while standing, handling a wheelchair, client bathing, client dressing, and housekeeping tasks. All items were assessed on the same frequency scale of almost never, about 25% of the time, about half of the time, about 75% of the time, and almost always

SECONDARY OUTCOMES:
Change from baseline in blood pressure at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Direct measurement via Omron HEM-907 automatic blood pressure monitor.
Change from baseline in blood lipids at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Direct measurement of total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides via Cholestech LDX Analyzer.
Change from baseline in blood glucose at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Direct measurement via Cholestech LDX Analyzer
Change from baseline in body weight at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Direct measurement via Tanita TBF-310GS Bioelectric Impedance Analyzer.
Change from baseline in body mass index (BMI) at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Direct measurement of height via SECA 213 portable stadiometer. Direct measurement of weight via Tanita TBF-310GS Bioelectric Impedance Analyzer. Calculation of BMI using direct measurements of height and weight.
Change from baseline in percent body fat at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Direct measurement via Tanita TBF-310GS Bioelectric Impedance Analyzer.
Change from baseline in body measurements at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Direct measurement of neck, waist, and hip circumference via Gulick II measuring tape. Calculation of waist hip ratio.
Change from baseline in stress at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Survey measures: Stress In General (Stanton et al., 2001), Interpersonal Conflict (Wright et al., 2014), Perceived Stress (Cohen et al., 1983).
Change from baseline in sleep quality and fatigue at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Survey measures: Single item from the Pittsburgh Sleep Quality Index (Buysse et al., 1989), Swedish Occupational Fatigue Inventory (Ahsberg, 2000)
Change from baseline in social support at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Survey measures: Social Support for Diet Behaviors (Sallis et al., 1987), Social Support for Exercise Behaviors (Sallis et al., 1987), Social Support Network (Toseland, 1990).
Change from baseline in musculoskeletal symptoms at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Survey measures: Adapted Nordic Questionnaire for Musculoskeletal Symptoms and functional impairment with activities of daily living (Dennerlein et al., 2012).
Change from baseline in illnesses and injuries at 6 and 12 months. Post intervention maintenance from 12 to 24 months. | Baseline, 6 months, 12 months, 24 months
  Survey measures: Self-reported lost time and first aid injuries, self-reported diagnoses of and treatment for co-morbid conditions.
Change from baseline in grip strength at 6 and 12 months. Post intervention maintenance from 12 to 24 months | Baseline, 6 months, 12 months, 24 months
  Measure: Grip strength (kg)
Change from baseline in hamstring flexibility at 6 and 12 months. Post intervention maintenance from 12 to 24 months | Baseline, 6 months, 12 months, 24 months
  Measure: Hamstring flexibility (in)
Change from baseline in 6-minute walk test at 6 and 12 months. Post intervention maintenance from 12 to 24 months | Baseline, 6 months, 12 months, 24 months
  Measure: Walking distance in six minutes (meters)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Olson R, Wright RR, Elliot DL, Hess JA, Thompson S, Buckmaster A, Luther K, Wipfli B. The COMPASS pilot study: a total worker Health intervention for home care workers. J Occup Environ Med. 2015 Apr;57(4):406-16. doi: 10.1097/JOM.0000000000000374. PMID 25654631
- [Background] Olson R, Elliot D, Hess J, Thompson S, Luther K, Wipfli B, Wright R, Buckmaster AM. The COMmunity of Practice And Safety Support (COMPASS) Total Worker Health study among home care workers: study protocol for a randomized controlled trial. Trials. 2014 Oct 27;15:411. doi: 10.1186/1745-6215-15-411. PMID 25348013
- [Background] Olson R, Elliot DL, Hess JA, Thompson S, Luther K, Wipfli B. COMPASS: Protecting and promoting the health of direct care givers. California Association for Behavior Analysis Western Regional Conference, San Diego, CA. February 2015.
- [Background] Olson R, Elliot DL, Hess JA, Thompson S, Wright RR, Luther K, Mancini A, Wipfli B. COMPASS teams: Creating health & safety "communities of practice" for home care workers. Teaming up for Total Worker Health symposium at the NIOSH 1st International Symposium to Advance Total Worker Health, Bethesda, MD. October 2014.
- [Background] Olson R, Thompson S, Hess JA. A Total Worker Health program for health care workers. National HealthCare Ergonomics Conference, Portland, OR. September 2014.
- [Background] Olson R, Wright R, Elliot DE, Hess J, Wipfli B, Mancini A. The COMPASS Pilot Study: A Total Worker Health Intervention for Home Care Workers. International Work, Stress, and Health conference, Los Angeles, CA. May 2013.
- [Background] Olson R, Thompson S. Behavior change tactics you can apply today: Findings and tools from the COMPASS total worker health program for home care workers. Oregon Governor's Occupational Safety & Health conference, Portland, OR. March 2015.
- [Background] Olson R. A Total Worker Health program for home care workers: Six month outcomes. UW/ UBC/ SFU/ Uvic/OSU Annual Conference on Environmental, Occupational, and Population Health, Semiahmoo Resort, WA. January 2015
- See also: Related Info — http://www.ohsu.edu/xd/research/centers-institutes/oregon-institute-occupational-health-sciences/oregon-healthy-workforce-center/projects/compass/